CLINICAL TRIAL: NCT01447173
Title: Vitamin and Asthma Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Yanbin Dong, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VDAS
Record Dates: First submitted 2011-10-03; First posted 2011-10-06 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: Asthma; Pulmonary Function Test; Vitamin D
MeSH Terms: conditions — Asthma | interventions — Vitamin D

ARMS (2):
- 2000 IU vitamin D Daily (Experimental)
  Interventions: Drug: Vitamin D
- 400 IU Vitamin D pill (Placebo Comparator)
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D 2000 IU daily pill Vitamin D 400 IU daily pill

SUMMARY:
The study looks at how vitamin D supplement will improve the severity of asthma and lung function as well as biomarkers in asthmatic children.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma (under control)otherwise in good general health

Exclusion Criteria:

* Poorly controlled asthma
* Taking daily multivitamin or vitamin D supplementation
* Taking oral steroid medication
* History of bronchopulmonary dysplasia or chronic lung disease, extreme prematurity, congenital heart disease, significant renal dysfunction or primary kidney disease, endocrinologic abnormalities of calcium metabolism or parathyroid disorders

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Function Test (PFT) after vitamin D supplementation | 4 weeks
Change in Asthma Control Test (ACT) scores after vitamin D supplementation | 4-week

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatrics Allergy Clinic at Georgia Health Sciences University, Augusta, Georgia, United States